CLINICAL TRIAL: NCT02350764
Title: An Exploratory Study to Evaluate the Mediators of Sensitivity and Resistance to Nivolumab Plus Ipilimumab in Patients With Advanced NSCLCs
Brief Title: Evaluate the Mediators of Sensitivity and Resistance to Nivolumab Plus Ipilimumab in Patients With Advanced NSCLCs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-137
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2023-09

CONDITIONS: Advanced Stage Non-small Cell Lung Cancer
Keywords: Nivolumab; Lung; ipilimumab; NSCLC; 14-137
MeSH Terms: interventions — Nivolumab

ARMS (1):
- Nivolumab (Experimental): Patients will begin treatment with nivolumab IV 3mg/kg and ipilimumab 1mg/kg. Treatment with nivolumab will continue every 2 weeks (+/- 3 days) thereafter and treatment with ipilimumab will continue every 6 weeks (+/- 3 days) thereafter. Treatment will continue until protocol-defined toxicity, confirmed progression of disease*, withdrawal of consent, or death.
  Interventions: Drug: nivolumab; Drug: pilimumab

INTERVENTIONS:
Drug: nivolumab
Drug: pilimumab

SUMMARY:
The purpose of this study is to closely examine tumor and blood samples from patients treated with nivolumab and ipilimumab in order to try to identify why some patients with lung cancers respond and why some patients do not.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be capable, willing, and able to provide written, informed consent.
* ≥ 18 years old.
* Advanced stage NSCLC
* Previously treated with no more than two lines of prior systemic therapy for advanced stage lung cancer.

  * Patients who previously received neoadjuvant, concurrent, or adjuvant chemotherapy for localized NSCLC and then recurred within 6 months of completing chemotherapy may be considered as having received one line of prior therapy
  * Maintenance therapy does not count as a separate line of therapy
* Patients must:

  * Be scheduled to undergo a standard-of-care resection of tumor tissue as part of treatment plan prior to beginning study therapy. Patients may not have intervening systemic anti-cancer therapy between the time of resection and treatment with nivolumab.
  * Have collection of adequate pre-treatment tissue for correlative analysis defined as sufficient material for 1) frozen tissue for DNA/RNA with touch prep/representative slide confirming tumor material present, 2) FFPE material for ICH with touch prep/representative slide confirming tumor material present, and 3) single-cell suspensions with >20 million live cells after tissue digestion but before freezing. Adequacy of collected material will be determined within 5 business days of each collected case.
  * Have residual disease following surgical resection that is measurable by RECIST v1.1
  * Previously irradiated sites of tumor may be considered measurable if there is radiographic progression at that site subsequent to the time of completing radiation.
  * Have a safely biopsiable tumor lesion
* ECOG performance status of 0-1.
* Adequate hematologic, renal, and/or hepatic function (following criteria must be met within 28 days of C1D1:

  * WBC ≥ 2,000/ul
  * ANC ≥ 1,500/ul
  * Hemoglobin ≥ 9.0 g/dl
  * Platelet count ≥ 100,000/ul
  * Total bilirubin ≤ 1.5 x ULN (unless evidence of Gilbert's syndrome, in which case, direct bilirubin must be ≤ 1.0 x ULN)
  * AST and ALT ≤ 3 x UNL (unless elevated transaminases are felt to be directly related to metastatic disease involving the liver, in which case AST and ALT must be ≤ 5x ULN)
  * Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance of ≥ 40 mL/min calculated using the formula of Cockcroft and Gault: (140-Age) • Mass (kg)/(72 • creatinine mg/dL); multiply by 0.85 if female
* There is no restriction on the number of prior lines of systemic anti-cancer therapy. For those who have received prior systemic anti-cancer therapy, there must be at least 3 weeks since last systemic therapy.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 3 days prior to the start of study drug.
* Effective contraception:

  * Women of childbearing potential must agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 23 weeks (5 half-lifes plus 30 days, the duration of an ovulatory cycle) after the last dose of nivolumab, or agree to completely abstain from heterosexual intercourse.
  * Male subjects, even if surgically sterilized (i.e., status post vasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through 31 weeks (5 half-lives plus 90 days, the duration of sperm turnover) after the last dose of study drug, or completely abstain from heterosexual intercourse.

Exclusion Criteria:

* Patients who are pregnant or lactating.
* Presence of activating EGFR mutations or ALK re-arrangement,unless previously treated with standard TKI therapy. All patients with adenocarcinoma histology must be tested for EGFR and ALK status.
* History of allergy to study drug components or history of severe hypersensitivity reaction of any monoclonal antibody.
* Prior treatment with immune checkpoint inhibitor, including (but not limited to) those targeting PD-1, PD-L1, PD-L2, CTLA-4, CD137, GITR, TIM3, LAG3, or OX40
* Any systemic anti-cancer therapy within 3 weeks prior to C1D1 of study therapy
* Exception is made for patients with EGFR or ALK re-arrangements who must have stopped TKI therapy at least 7 days prior to C1D1
* Patients who have not previously been treated with platinum-based based doublet chemotherapy and who, in the judgment of the investigator, have rapidly progressive disease such that serious complications may arise from disease progression within the next 12 weeks will be excluded.
* Non-CNS radiotherapy within 1 week prior to C1D1 of study therapy
* Active infection requiring therapy
* Prior systemic immunosuppressive therapy (> 10 mg/day prednisone equivalents) within 1 week prior to C1D1 of study therapy. Inhaled, ocular, intra-articular, intranasal, and topical corticosteroids are permitted in absence of active autoimmune disease.

  * Adrenal replacement doses are permitted in the absence of active autoimmune disease.
* Patients with known or suspected history of autoimmune disease. Subjects with type I diabetes melitis, hypothyroidism only requiring hormone replacement, resolved childhood asthma/atopy, patients with asthma requiring intermittent bronchodilator therapy, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Other active malignancy requiring concurrent intervention.
* Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, cervical/dysplasia, melanoma, or breast) are excluded unless definitive therapy has been completed at least 1 year prior to study entry and the patient is now without evidence of disease from that malignance and no additional therapy is required or anticipated to be required during the study period.
* Known untreated brain or leptomeningeal metastasis.

  o Patients with brain metastases are eligible if metastases have been adequately treated and neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least two weeks prior to C1D1. In addition, must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
* Patients with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Any positive test for HIV
* Any positive test for HCV RNA or HBsAg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Schoenfeld, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab: Patients will begin treatment with nivolumab IV 3mg/kg and ipilimumab 1mg/kg. Treatment with nivolumab will continue every 2 weeks (+/- 3 days) thereafter and treatment with ipilimumab will continue every 6 weeks (+/- 3 days) thereafter. Treatment will continue until protocol-defined toxicity, confirmed progression of disease*, withdrawal of consent, or death.
  nivolumab
  pilimumab
Period: Overall Study
Arm/Group | Nivolumab
Started | 29
Completed | 18
Not Completed | 11
Not completed — Adverse Event | 4
Not completed — Death | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab
Number analyzed (Participants) | 29
Age, Continuous [Mean (Full Range); unit: years] | 61.9 [44.9 to 81.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (Confirmed Partial + Complete Response) Will be Assessed as Part of This Study. Tumor Response Will be Assessed Using RECIST 1.1)
Description: confirmed partial + complete response will be assessed as part of this study. Tumor response will be assessed using RECIST 1.1. All responses must be confirmed on subsequent scan to be considered a true response. Tumor assessments will be performed after.6 weeks (+/- 1 week) and subsequently every six week (+/- 1 week) thereafter while on study until week 48. After week 48, tumor assessments will be conducted every 12 weeks (+/- week). Additional tumor assessments may be performed at the discretion of the treating physician.
Time Frame: every 6 weeks (+/- 1 week) until week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab
Number analyzed (Participants) | 29
Participants
  Stable Disease | 7
  Progression of Disease | 5
  Partial Response | 5
  Not entered | 12

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Nivolumab
All-Cause Mortality (participants affected / at risk) | 14/29
Serious Adverse Events (participants affected / at risk) | 22/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=29)
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 3
Fatigue (General disorders) | 1
Neck edema (General disorders) | 1
Abdominal infection (Infections and infestations) | 1
Bronchial infection (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pleural infection (Infections and infestations) | 1
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Neoplasms ben/mal/unk (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Seizure (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=29)
Hyperglycemia (Metabolism and nutrition disorders) | 29
Hypoalbuminemia (Metabolism and nutrition disorders) | 27
Anemia (Blood and lymphatic system disorders) | 22
Hypomagnesemia (Metabolism and nutrition disorders) | 19
Alkaline phosphatase increased (Investigations) | 17
Fatigue (General disorders) | 17
Hyponatremia (Metabolism and nutrition disorders) | 17
Hypocalcemia (Metabolism and nutrition disorders) | 16
Lymphocyte count decreased (Investigations) | 15
Platelet count decreased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 13
Hypokalemia (Metabolism and nutrition disorders) | 13
Alanine aminotransferase increased (Investigations) | 13
Constipation (Gastrointestinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13
INR increased (Investigations) | 11
Anorexia (Metabolism and nutrition disorders) | 11
Pain (General disorders) | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8
Nausea (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 8
Activated partial thromboplastin time prolonged (Investigations) | 8
White blood cell decreased (Investigations) | 8
Serum amylase increased (Investigations) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 6
Weight loss (Investigations) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 6
Edema limbs (General disorders) | 6
Anxiety (Psychiatric disorders) | 5
Lipase increased (Investigations) | 5
Myalgia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Creatinine increased (Investigations) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Paresthesia (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 5
Blood bilirubin increased (Investigations) | 4
Lung infection (Infections and infestations) | 4
Cholesterol high (Investigations) | 4
Depression (Psychiatric disorders) | 4
Skin infection (Infections and infestations) | 4
Hyperthyroidism (Endocrine disorders) | 4
Fever (General disorders) | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 3
Non-cardiac chest pain (General disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Hot flashes (Vascular disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Headache (Nervous system disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 3
Thromboembolic event (Vascular disorders) | 3
Hypertension (Vascular disorders) | 3
Hypothyroidism (Endocrine disorders) | 3
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
Upper respiratory infection (Infections and infestations) | 2
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 2
Seizure (Nervous system disorders) | 2
Watering eyes (Eye disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Dry eye (Eye disorders) | 2
Hemoglobin increased (Investigations) | 2
Hypotension (Vascular disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Palpitations (Cardiac disorders) | 2
Urinary frequency (Renal and urinary disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Neutrophil count decreased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT02350764/Prot_SAP_000.pdf